CLINICAL TRIAL: NCT00059410
Title: Alzheimer's Disease Treatment and Illness Perceptions Survey (TIPS) II
Status: Completed | Type: Observational
Sponsor: Alzheimer's Association (Other)
Organization: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0045; NIRG-02-3712; BUMC 2002-308
Record Dates: First submitted 2003-04-24; First posted 2003-04-28 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Caregivers; African Americans; Perceptions; Cultural Competency
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The TIPS Study, or Treatment and Illness Perceptions Survey, is a study funded by the national Alzheimer's Association to learn more about differences between African Americans' and Whites' attitudes, beliefs, and experiences related to Alzheimer's disease (AD). The study involves a one-time 30-minute telephone survey in which participants are asked about a range of topics related to AD, including their personal experiences, their beliefs about the disease's symptoms and risk factors, and their attitude toward possible future treatment options. Information from the survey will be used to develop more culturally sensitive health education and healthcare services for persons with AD.

DETAILED DESCRIPTION:
The main goal of the Boston University's TIPS II project is to examine differences in Alzheimer's disease (AD) illness perceptions between African Americans and Whites in order to better understand attitudes and beliefs and to develop more culturally sensitive health services for AD. This 30-minute telephone survey will include a total of 140 first-degree relatives and caregivers of people with AD, as well as a comparison group of 70 adults without family history. The researchers will assess 1) beliefs about AD; 2) the perceived threat it poses; 3) sources of information about AD; 4) knowledge of basic facts about AD; 5) appraisal of AD treatments; and 6) intentions regarding current and emerging care options. Based on preliminary data, this study hypothesize that, as compared to Whites, African Americans will report lower levels of perceived threat, fewer sources of information, less awareness of facts, and less interest in care options. Focus group interviews with African American participants will help interpret study findings and inform recommendations for health education interventions.

Findings will inform the development of a set of recommendations for AD health educators that will help them tailor their interventions to African Americans. Such educational programs promote increased use of assessment, treatment, and caregiver assistance services. Results will also be used as pilot data in a proposal for a national survey of caregivers and relatives. This program of research will address a growing need for increased understanding of beliefs, knowledge, and intentions regarding AD. A total of 210 participants are being sought (105 African Americans, and 105 Whites). Participants who complete the survey will be given a $10.00 check, plus informational brochures on AD and the latest newsletter from the Boston University Alzheimer's Disease Center.

ELIGIBILITY:
Inclusion Criteria:

Three groups of participants are sought to take part in the survey:

* 70 primary caregivers(current or former) of persons with AD, or related memory disorders
* 70 adult children and siblings of people with AD or related memory disorders
* 70 adults age 40 and older without immediate family history of AD or related memory disorders

Exclusion Criteria:

* Not fluent in English
* Cognitive impairment that would preclude responding to a 30-minute telephone survey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2003-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Roberts, PhD, Study Director — Boston University Alzheimer's Disease Center
Locations (1):
- Boston University School of Medicine, Alzheimer's Disease Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Roberts JS, Connell CM. Illness representations among first-degree relatives of people with Alzheimer disease. Alzheimer Dis Assoc Disord. 2000 Jul-Sep;14(3):129-136,Discussion 127-8. doi: 10.1097/00002093-200007000-00003. PMID 10994653
- [Background] Roberts JS. Anticipating response to predictive genetic testing for Alzheimer's disease: a survey of first-degree relatives. Gerontologist. 2000 Feb;40(1):43-52. doi: 10.1093/geront/40.1.43. PMID 10750312
- [Background] Roberts JS, Connell CM, Cisewski D, Hipps YG, Demissie S, Green RC. Differences between African Americans and whites in their perceptions of Alzheimer disease. Alzheimer Dis Assoc Disord. 2003 Jan-Mar;17(1):19-26. doi: 10.1097/00002093-200301000-00003. PMID 12621316